CLINICAL TRIAL: NCT06220396
Title: CArdioMEtabolic Function and Reserve Capacity in Healthy Adults: The CAMERA Study
Acronym: CAMERA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Barry Borlaug, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 23-007522
Record Dates: First submitted 2023-12-28; First posted 2024-01-23 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Healthy
MeSH Terms: interventions — Hemodynamics; Magnetic Resonance Spectroscopy; Absorptiometry, Photon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Volunteers (Experimental): Healthy volunteers with no history of Heart Failure (HF) will undergo a Right Heart Catheterization with Hemodynamics and Limited Echocardiogram, MRI, and DEXA scan.
  Interventions: Procedure: Right Heart Catheterization with Hemodynamics and Limited Echocardiogram; Procedure: Magnetic Resonance Imaging (MRI); Procedure: Dual X-ray absorptiometry (DEXA) scan

INTERVENTIONS:
Procedure: Right Heart Catheterization with Hemodynamics and Limited Echocardiogram — Right Heart Catheterization (RHC) with Hemodynamics and Limited Echocardiogram is an invasive procedure that involves insertion of a catheter through a blood vessel in the neck, groin, or arm to the right side of the heart. Hemodynamic measurements such as the blood pressure inside the veins, heart, and arteries as well as measurements of blood flow and how much oxygen is in the blood will be completed during the catheterization procedure. It is a way to see how well the heart is working during your procedure. During the RHC procedure a limited echocardiogram, using ultrasound waves, will be collected to evaluate the structure and function of the heart.
  All measurements will be conducted at rest and during exercise using a supine cycle ergometer
Procedure: Magnetic Resonance Imaging (MRI) — MRI is a medical imaging technique that uses a magnetic field and computer-generated radio waves to create detailed images of the organs and tissues in your body. CMR Imaging will assess myocardial structure, function, and fat content.
  An additional limited MRI sequence of the the abdomen and one sequence in the thigh will be used to evaluate for visceral adipose tissue (VAT) as a measurement of body composition.
  Other Names: CMR Imaging
Procedure: Dual X-ray absorptiometry (DEXA) scan — A DEXA scan measures the amount of fat in the body using an x-ray that measures bone, calcium and fat.

SUMMARY:
The purpose of this study is to evaluate pulmonary capillary wedge pressure (PCWP) and other hemodynamic measurements at rest and during exercise in healthy volunteers across the age spectrum.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy volunteers are eligible to participate in this study if they are free of symptoms of exertional breathlessness or fatigue and any diagnosis of heart failure.
* Patients will also be required to have left ventricular ejection fraction (EF) ≥ 50%.
* Patients discovered to reduced EF or abnormal resting hemodynamics or other pathologic findings previously undiscovered will be considered screen failures and can be replaced by others to reach the goal enrollment.
* Informed consent were obtained.
* No history of heart failure.
* Willing and able to undergo invasive hemodynamic exercise testing, MRI, and other study assessments.

Exclusion Criteria:

* Clinically significant symptoms of exertional dyspnea or fatigue in daily life in the opinion of the investigators.
* Any diagnosis of heart failure
* Symptomatic coronary artery disease (e.g., patients with chronic angina)
* Symptomatic valvular heart disease
* Pulmonary hypertension
* Cardiomyopathies
* High output heart failure
* Pericardial disease
* Clinically significant chronic lung disease in the opinion of the investigators
* Anemia (hemoglobin <12 gm/dL in women and <13 gm/dL in men)
* Estimated glomerular filtration rate ≤30mL/min
* Pregnant women
* Any other disorders or problems that would interfere with the ability to participate safely in the study (e.g. psychiatric disorder or substance abuse)

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Capillary Wedge Pressure (PCWP) at rest | Baseline
  Pulmonary capillary wedge pressure is a measure of cardiac filling pressure, measured using a high-fidelity micromanometer advanced through the lumen of a fluid-filled catheter at rest.
Pulmonary Capillary Wedge Pressure (PCWP) during exercise | Baseline
  Pulmonary capillary wedge pressure is a measure of cardiac filling pressure, measured using a high-fidelity micromanometer advanced through the lumen of a fluid-filled catheter during exercise.

SECONDARY OUTCOMES:
Trans-cardiac uptake of free fatty acids (FFA) at rest | Baseline
  Trans-cardiac uptake of FFA will be measured using arterial and coronary sinus blood samples collected at rest during cardiac catheterization procedure.
Trans-cardiac uptake of free fatty acids (FFA) during exercise | Baseline
  Trans-cardiac uptake of FFA will be measured using arterial and coronary sinus blood samples collected during the exercise portion of the cardiac catheterization procedure.
Trans-cardiac uptake of glucose at rest | Baseline
  Trans-cardiac uptake of glucose will be measured using arterial and coronary sinus blood samples collected at rest during the cardiac catheterization procedure.
Trans-cardiac uptake of glucose during exercise | Baseline
  Trans-cardiac uptake of glucose will be measured using arterial and coronary sinus blood samples collected during the exercise portion of the cardiac catheterization procedure.
Trans-cardiac uptake of ketone bodies at rest | Baseline
  Trans-cardiac uptake of ketone bodies will be measured using arterial and coronary sinus blood samples collected at rest during the cardiac catheterization procedure.
Trans-cardiac uptake of ketone bodies during exercise | Baseline
  Trans-cardiac uptake of ketone bodies will be measured using arterial and coronary sinus blood samples collected during the exercise portion of the cardiac catheterization procedure.
Left ventricular (LV) global longitudinal strain | Baseline
  LV global longitudinal strain will be assessed by echocardiography conducted during the cardiac catheterization procedure
Left Atrial (LA) reservoir strain | Baseline
  LA reservoir strain will be assessed by echocardiography conducted during the cardiac catheterization procedure
Right Ventricular (RV) free wall strain | Baseline
  RV free wall strain will be assessed by echocardiography conducted during the cardiac catheterization procedure
Myocardial mass | Baseline
  Myocardial mass will be measured by CMR imaging.
Myocardial volume | Baseline
  Myocardial volume will be measured by CMR imaging.
Myocardial fat content | Baseline
  Myocardial fat content will be measured by CMR imaging.
Body fat mass | Baseline
  Body fat mass will be measured using dual X-ray absorptiometry (DEXA)
Visceral fat content | Baseline
  Visceral fat content will be measured using limited abdominal MRI
Total blood volume | Baseline
  Total blood volume will be assessed by using the radiolabeled iodinated albumin (131I, 5-25 μCu) indicator dilution technique (BVA-100 Blood Volume Analyzer, Daxor Corp, NY).
Total plasma volume | Baseline
  Total plasma volume will be assessed by using the radiolabeled iodinated albumin (131I, 5-25 μCu) indicator dilution technique (BVA-100 Blood Volume Analyzer, Daxor Corp, NY).
Quality of Life (QOL) as assessed by Kansas City Cardiomyopathy Questionnaire (KCCQ) | Baseline
  KCCQ was a 23-item, self-administered questionnaire that measure the participant's perception of their health status, including their heart failure (HF) symptoms, impact on physical and social function and how their HF impacts the quality of life. KCCQ quantifies 7 domains: physical limitations (6 items), symptom stability (1 item), symptom frequency (4 items), symptom burden (3 items), self-efficacy (2 items), quality of life (3 items) and social limitations (4 items). Scores were generated for each domain and scaled from 0 to 100, with 0 (worst) and 100 (the best possible status), where the higher score reflected better health status.
Blood glucose level | Baseline
  Blood glucose level will be measured using oral glucose tolerance testing
Blood insulin level | Baseline
  Blood insulin level will be measured using oral glucose tolerance testing
Blood free fatty acids (FFA) level | Baseline
  Blood FFA level will be measured using oral glucose tolerance testing

CONTACTS AND LOCATIONS:
Overall Officials: Barry Borlaug, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No